CLINICAL TRIAL: NCT02596451
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence of Diclofenac Sodium Gel, 1% (Glenmark Pharmaceuticals Ltd) to Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% (Novartis Consumer Health, Inc) in Patients With Osteoarthritis (OA) of the Knee
Brief Title: To Study Generic Diclofenac Sodium Topical Gel 1% in the Treatment of Osteoarthritis of the Knee (Degenerative Joint Disease Presented as Joint Pain, Stiffness, Swelling and Restricted Motion).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLK-1402
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2016-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac Sodium gel, 1% (Experimental): apply gel to the target knee
  Interventions: Drug: Diclofenac Sodium gel, 1%
- Voltaren® Gel (Active Comparator): apply gel to the target knee
  Interventions: Drug: Voltaren® Gel
- Placebo (Placebo Comparator): apply gel to the target knee
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac Sodium gel, 1%
  Arms: Diclofenac Sodium gel, 1%
Drug: Voltaren® Gel
  Arms: Voltaren® Gel
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence of Diclofenac Sodium Gel, 1% (Glenmark Pharmaceuticals Ltd) to Voltaren® Gel (Diclofenac Sodium topical gel) 1% (Novartis Consumer Health, Inc) in Patients with Osteoarthritis (OA) of the Knee

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female aged ≥ 35 years with a clinical diagnosis of OA of the knee according to the American College of Rheumatology (ACR) criteria.
2. OA Symptoms for at least 6 months prior to screening.
3. Baseline Western Ontario McMaster Osteoarthritis (WOMAC) pain subscale of > 9 on a 20 point scale for the target knee immediately prior to randomization.

Exclusion Criteria:

1. History of OA pain in the contralateral knee requiring medication within 1 year prior to screening.
2. History of secondary OA, rheumatoid arthritis, chronic inflammatory disease (e.g., colitis) or fibromyalgia.
3. History of gastrointestinal bleeding or peptic ulcer disease.
4. Known allergy to aspirin or nonsteroidal anti-inflammatory drug (NSAID).
5. Use of anticoagulants, ACE-inhibitors, cyclosporine, diuretics, lithium, or methotrexate prior to 30 days of screening.
6. Concomitant use of systemic corticosteroids, topical corticosteroids, or immunosuppressive drugs or their use prior to 30 days of screening.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh V Deshpande, Study Director — Glenmark Pharmaceuticals Ltd
Locations (44):
- United States (44):
  - Glenmark Investigational Site 5, Mesa, Arizona
  - Glenmark Investigational Site 1, Anaheim, California
  - Glenmark Investigational Site 21, Anaheim, California
  - Glenmark Investigational Site 31, Anaheim, California
  - Glenmark Investigational Site 26, Canoga Park, California
  - Glenmark Investigational Site 42, Carlsbad, California
  - Glenmark Investigational Site 30, Carmichael, California
  - Glenmark Investigational Site 33, Cerritos, California
  - Glenmark Investigational Site 25, El Cajon, California
  - Glenmark Investigational Site 24, La Mesa, California
  - Glenmark Investigational Site 2, Pasadena, California
  - Glenmark Investigational Site 13, Rancho Cucamonga, California
  - Glenmark Investigational Site 27, Sacramento, California
  - Glenmark Investigational Site 10, Fort Lauderdale, Florida
  - Glenmark Investigational Site 41, Hialeah, Florida
  - Glenmark Investigational Site 15, Miami, Florida
  - Glenmark Investigational Site 19, Miami, Florida
  - Glenmark Investigational Site 28, Miami, Florida
  - Glenmark Investigational Site 32, Miami, Florida
  - Glenmark Investigational Site 40, Miami, Florida
  - Glenmark Investigational Site 3, Miami Lakes, Florida
  - Glenmark Investigational Site 37, Ormond Beach, Florida
  - Glenmark Investigational Site 11, West Palm Beach, Florida
  - Glenmark Investigational Site 18, West Palm Beach, Florida
  - Glenmark Investigational Site 8, Evanston, Illinois
  - Glenmark Investigational Site 43, Newburgh, Indiana
  - Glenmark Investigational Site 38, Wichita, Kansas
  - Glenmark Investigational Site 17, New Orleans, Louisiana
  - Glenmark Investigational Site 22, Saginaw, Michigan
  - Glenmark Investigational Site 14, St Louis, Missouri
  - Glenmark Investigational Site 9, Englewood, Ohio
  - Glenmark Investigational Site7, Altoona, Pennsylvania
  - Glenmark Investigational Site 36, Knoxville, Tennessee
  - Glenmark Investigational Site 39, Nashville, Tennessee
  - Glenmark Investigational Site 23, Beaumont, Texas
  - Glenmark Investigational Site 20, Bryan, Texas
  - Glenmark Investigational Site 34, Dallas, Texas
  - Glenmark Investigational Site 35, Houston, Texas
  - Glenmark Investigational Site 44, Houston, Texas
  - Glenmark Investigational Site 4, Lampasas, Texas
  - Glenmark Investigational Site 29, San Antonio, Texas
  - Glenmark Investigational Site 6, San Antonio, Texas
  - Glenmark Investigational Site 16, Charlottesville, Virginia
  - Glenmark Investigational Site12, Midlothian, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Test: Diclofenac Sodium gel, 1% (Glenmark Pharmaceuticals Ltd)
- Reference: Voltaren® Gel (Diclofenac Sodium topical gel) 1% (Novartis Consumer Health, Inc)
- Placebo: Vehicle gel (Glenmark Pharmaceuticals Ltd)
Period: Overall Study
Arm/Group | Test | Reference | Placebo
Started | 385 | 392 | 387
Completed | 381 | 374 | 373
Not Completed | 4 | 18 | 14

BASELINE CHARACTERISTICS:
Population: A total of 1164 subjects were randomized in the study; however there were 21 subjects excluded from the safety population randomized who did not received dose. (Test=2, Reference=10, Placebo=9). Therefore the subject numbers are not consistent with any of the rows in the Participant Flow module.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Placebo | Total
Number analyzed (Participants) | 383 | 382 | 378 | 1143
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.36) | 56.5 (10.68) | 56.7 (10.52) | 56.4 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 237 | 248 | 734
  Male | 134 | 145 | 130 | 409

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in the Total WOMAC (Western Ontario and McMaster Universities Arthritis Index) Pain Subscale Score for the Target Knee
Description: The total WOMAC Pain Subscale score was determined by summing the individual scores from each of the five questions using a 5-point Likert scale (i.e., 'none'=0; 'mild'=1, 'moderate'=2; 'severe'=3; 'extreme'=4) comprising the WOMAC Pain Subscale Rating for the Target Knee.
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test | Reference
Number analyzed (Participants) | 309 | 285
units on a scale | 5.8 (3.96) | 5.9 (3.94)

ADVERSE EVENTS:
Arm/Group | Test | Reference | Placebo
Serious Adverse Events (participants affected / at risk) | 0/383 | 2/382 | 1/378
Other Adverse Events (participants affected / at risk) | 28/383 | 26/382 | 23/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=383) | Reference (N=382) | Placebo (N=378)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
L Ankle Surgery Secondary To Trimalleolar Fracture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Right Ankle Surgery Due To Stair Fall (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) — This SAE was occured during the baseline lead-in period of the study and subject did not use the study product.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=383) | Reference (N=382) | Placebo (N=378)
Headache (Nervous system disorders) | 28 (38) | 26 (46) | 23 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the agreement, Sponsor reserves the right for publishing trial results and the Investigator cannot publish without written consent from the Sponsor.